CLINICAL TRIAL: NCT03233061
Title: Does Obesity Influence Women Cardiorespiratory Fitness and Daily Physical Activities?
Brief Title: Does Obesity Influence Women Cardiorespiratory Fitness and Daily Physical Activities? (ACTIVOB)
Acronym: ACTIVOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratory of Movement, Condorcet, Tournai, Belgium (Other)
Responsible Party: Principal Investigator, Grégory Cuvelier, Laboratory Head, Laboratory of Movement, Condorcet, Tournai, Belgium
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017001
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: Obesity; cardiorespiratory fitness; oxygen uptake; household activities; physical activity; sedentary; intensity; obese women
MeSH Terms: conditions — Obesity; Motor Activity; Sedentary Behavior | interventions — Cardiorespiratory Fitness

STUDY DESIGN:
Intervention Model Description: Women OBESE group VS Women NON-OBESE group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NO (Active Comparator): NON OBESE WOMEN GROUP ( same age and same physical activities ) cardiorespiratory exercise testing with evaluation of peak oxygen uptake, heart rate and maximal cycling power output. Cardiorespiratory functioning is assessed during household activities such as ironing,cleaning floor,walking and climbing stairs.
  Interventions: Diagnostic Test: cardiorespiratory fitness and daily physical activities evaluations
- OB (Experimental): OBESE GROUP cardiorespiratory exercise testing with evaluation of peak oxygen uptake,heart rate and maximal cycling power output.Cardiorespiratory functioning is assessed during household activities such as ironing, cleaning floor, walking and climbing stairs
  Interventions: Diagnostic Test: cardiorespiratory fitness and daily physical activities evaluations

INTERVENTIONS:
Diagnostic Test: cardiorespiratory fitness and daily physical activities evaluations — The cardiopulmonary exercise testing is performed on a cycle ergometer connected to cardiovascular and respiratory software. Subjects have a facemask, which collected respiratory and metabolic variables.An incremental exercise test is performed up to exhaustion. ⩒O2 is recorded and heart rate is averaged by an electrocardiogram system.
  Cardiopulmonary exercise testing during household activities Subjects have to perform 3 everyday life household activities: ironing,cleaning floor,walking and climbing stairs.A wearable ambulatory indirect metabolic system is used with Holter mode to record cardiorespiratory measures.Subjects have to breathe through the K4b2 facemask and turbine.

SUMMARY:
Many obese individuals experience difficulties in executing household activities. In this study, we investigate the cardiorespiratory fitness (CRF) of obese vs. non-obese women, and the impact of obesity on cardiorespiratory functioning during daily household activities.

DETAILED DESCRIPTION:
Methods: On 48 sedentary female subjects will be assessed by cardiorespiratory exercise testing with evaluation of peak oxygen uptake (⩒O2), heart rate (HR) and maximal cycling power output. Next, cardiorespiratory functioning will be assessed during household activities such as ironing (A1), cleaning floor (A2), walking and climbing stairs (A3).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI = weight in kilograms/(height in meters) x (height in meters)) as: healthy obese (OB group (OB); BMI between 30 to 39.9 kg.m-2; n = 20), and healthy non obese (NO group (NO); BMI between 18.5 to 24.9 kg.m-2; n = 28).

Exclusion Criteria:

* comorbidities (other than obesity) :

  1. history of systemic hypertension or antihypertensive medication, diabetes mellitus, cardiovascular or respiratory disease, systemic disease, smoking;
  2. any drugs;
  3. BMI >40 kg.m-2;
  4. having a regular physical activity.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Comparison of relative peak oxygen consumption between obese and non-obese women , mesured with indirect calorimetry | 2 months
  ⩒O2 peak comparison between OB vs NO women. For each household activity, the intensity expressed by the ratio ⩒O2 activity/resting ⩒O2 or the ratio ⩒O2 activity /⩒O2 peak will be compared between NO and OB

CONTACTS AND LOCATIONS:
Locations (1):
- LAboratoire de l'effort et du mouvement, Tournai, HAinaut, Belgium

IPD SHARING:
Plan to Share IPD: No